CLINICAL TRIAL: NCT01823172
Title: Feasibility of Lymphatic Mapping of Second Echelon Lymph Nodes With Methylene Blue
Brief Title: Second Echelon Node Study With Methylene Blue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James W. Jakub, Breast and Melanoma Surgery Section Head, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-009929
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer; Melanoma
Keywords: breast cancer; melanoma; sentinel lymph node biopsy; lymphadenectomy
MeSH Terms: conditions — Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylene Blue (Experimental): 1% Methylene Blue - 1 ml. Methylene blue dye injection of sentinel lymph node
  Interventions: Procedure: Methylene blue dye injection of sentinel lymph node

INTERVENTIONS:
Procedure: Methylene blue dye injection of sentinel lymph node — Single arm study. Methylene blue will be injected into the 1st SLN and traced via the efferent lymphatic to the 2nd echelon lymph node.

SUMMARY:
The investigators plan to study the ability to identify the lymph nodes beyond the sentinel lymph node that may harbor cancer using methylene blue dye.

DETAILED DESCRIPTION:
After lymphatic mapping of the SLN with Tc-99 sulfur colloid only, the second-echelon lymphatic mapping was then performed with methylene blue dye by injecting the SLN with 0.05-0.10 cc non dilute methylene blue and tracing via the efferent lymphatic channel to the second echelon lymph node (Figure 1). For our initial patients a 27 gauge needle and 3cc syringe was utilized but this was modified over the study to a 30 gauge needle and 1cc syringe. The blue efferent lymphatic was traced with minimal spreading of the surrounding tissue to visualize its drainage into the next lymph node(s). A second echelon lymph node was considered any blue lymph node or any lymph node with blue dye leading directly into it. The number of second echelon lymph nodes was recorded. The second-echelon lymph node(s) was not removed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary cutaneous melanoma located on the extremity or trunk
* Patients with clinically stage I-II melanoma
* Histologically confirmed invasive ductal or lobular carcinoma
* Patient undergoing surgical treatment of breast primary and sentinel lymph node biopsy- clinically node negative

Exclusion Criteria:

* Melanoma located on the head or neck, uveal or mucosal
* Previous surgery or radiation in or near the sentinel lymph node biopsy nodal basin
* Preoperative biopsy proven regional lymph node involvement
* Failure of lymphatic mapping with radioactive colloid
* Women who are pregnant or nursing
* Prior ipsilateral axillary surgery or radiation
* Inflammatory breast cancer
* No lymph node identified in the ipsilateral breast during pathologic review of the mastectomy specimen
* Stage IV breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The number of subjects in whom a secondary echelon lymph node is identified | one year

CONTACTS AND LOCATIONS:
Overall Officials: James Jakub, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share data